CLINICAL TRIAL: NCT00446888
Title: Effects of Nutritional Supplementation (Product 4808) on Acute Skeletal Muscle Protein Synthesis in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Robert R. Wolfe, PhD, UAMS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 71303
Record Dates: First submitted 2007-03-09; First posted 2007-03-13 (Estimated); Last update posted 2009-06-19 (Estimated); Status verified 2009-06

CONDITIONS: Cancer
Keywords: cancer; metastasis
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): these subjects will get a standard protein supplement "milkshake" during thei study.
  Interventions: Behavioral: Standardized Meals for Diet Stabilization; Dietary Supplement: Forticare
- 2 (Experimental): these subjects will receive an enhanced protein supplement "milkshake" during their study. Product 4808.
  Interventions: Behavioral: Standardized Meals for Diet Stabilization; Dietary Supplement: Product 4808

INTERVENTIONS:
Behavioral: Standardized Meals for Diet Stabilization — Subjects will eat prepared meals for 3 days prior to their study; or they will document their dietary intake over this period.
Dietary Supplement: Forticare — 400 ml of commercially-available nutritional supplement.
  Arms: 1
Dietary Supplement: Product 4808 — 400 ml Forticare, to which has been added extra protein and the amino acid leucine.
  Other Names: Product 4808.
  Arms: 2

SUMMARY:
The purpose of the study is to compare two different nutritional supplements with respect to their effect on building muscle, and to determine the factors that control the rate at which muscle tissue can be produced in subjects with cancer. After three days of receiving all meals from the Reynolds Institute on Aging in order to stabilize their diet, subjects will then return to the Institute to perform a single day study, where they will be given one of two supplements to drink. Blood will be taken from a catheter placed in one of their arms and three muscle biopsy samples will be taken from a leg. Subjects will have x-ray evidence of cancer and be 40 years of age or older in order to participate. It is the hypothesis that a nutritional supplement with a high amount of protein and containing leucine will target the metabolism problems in cancer patients.

DETAILED DESCRIPTION:
Muscle protein is generally diminished in cancer patients, with an effect on outcome. Research has shown that recurrence in treated patients is directly related to the extent of muscle loss. The effects of nutritional supplements; however, is still controversial. Anorexia due to metabolic changes in cancer patients can lead to reduced food intake and supplementation orally has often failed to show weight gain in these patients. These observations have led to the conclusion that even though food intake should be increased in order to gain lean body mass, this is difficult to achieve unless specific metabolic abnormalities are targeted.

This study is a comparison of two supplements on muscle protein synthesis. Approximately 40 patients with radiographic evidence of cancer, ages 40 and older will be enrolled.

Participation will require a screening procedure, including a history of medical problems and a physical exam, which may include blood testing for HIV or hepatitis as well as possibly for various basic diagnostic parameters. There may also be a urine-based drug screen or pregnancy test (if female). Participants should be in general good health and not have a variety of exclusion criteria.

There will be three days of diet stabilization, during which all meals will come from the Reynolds Institute of Aging. If subjects cannot comply with the diet, dietary recording will be substituted. Following these three days, there will be one day of main study activities. There will be catheters placed in both arms and blood samples will be taken from one of these. Stable amino acid isotopes will be infused into the bloodstream through the other. There will be three muscle biopsies taken from the thigh muscle throughout the day. Two doses of a nutritional supplements will be consumed 20 minutes apart during the main study day.

ELIGIBILITY:
Inclusion Criteria:

* radiographic evidence of Cancer
* Ages 40 and older
* Ability to sign Informed Consent

Exclusion Criteria:

* Patient received anti-cancer therapy or surgery less than 4 weeks prior to the experiment
* Body weight loss of more than 10% in past three months
* Body Mass Index less than 20kg/m2 or greater than 30 kg/m2
* Any documented autoimmune disease
* Peripheral vascular disease
* Hgb less than 9.0g/dL
* PT with INR greater than 1.5
* PTT greater than 40 seconds
* Platelet count less than 100,000
* Uncontrolled hypertension
* Currently using insulin to control high blood sugar
* Untreated metabolic diseases including liver or renal disease
* Currently in muscle strengthening program
* Use of supplements enriched with branched-chain amino acids
* History of hypo- or hyper-coagulation disorders, including patients taking Coumadin or history of deep venous thrombosis or pulmonary embolism at any point in their lifetime
* Currently taking aspirin and cannot stop for 7 days
* Presence of acute illness or metabolically unstable chronic illness
* Unstable heart disease requiring therapy or recent myocardial infarction (less than 1 year)
* Current alcohol or drug abuse
* Pregnancy or lactation (pre-menopausal women)
* Allergy/intolerance to any of the ingredients of the study products
* Any other condition deemed by the Principal Investigator and the study physician as exclusion or that interferes with proper study conduct or safety of the patient

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Muscle fractional synthetic rate of growth. | one day.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wolfe, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States